CLINICAL TRIAL: NCT01217944
Title: A 12 Month, Phase III, Randomized, Double-masked, Multicenter, Active-controlled Study to Evaluate the Efficacy and Safety of Two Different Dosing Regimens of 0.5 mg Ranibizumab vs. Verteporfin PDT in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia
Brief Title: Efficacy and Safety of Ranibizumab in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002F2301; 2010-021662-30 (EudraCT Number)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Pathological Myopia
Keywords: Pathologic myopia; PM; choroidal neovascularization; CNV; ranibizumab; verteporfin PDT
MeSH Terms: conditions — Myopia, Degenerative; Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Ranibizumab driven by disease activity (Experimental): Participants received active ranibizumab on day 1. Thereafter they received ranibizumab treatment based on disease activity criteria
  Interventions: Drug: Ranibizumab; Drug: Sham Ranibizumab; Drug: Sham verteporfin PDT
- Ranibizumab driven by stabilization criteria (Experimental): Participants received ranibizumab on day 1 and month 1. Thereafter they received ranibizumab based on stabilization criteria for visual acuity
  Interventions: Drug: Ranibizumab; Drug: Sham Ranibizumab; Drug: Sham verteporfin PDT
- Verteporfin PDT (Active Comparator): Participants received active vPDT on day 1. From month 3 onwards participants could receive ranibizumab, vPDT or a combination of the two if needed.
  Interventions: Drug: Ranibizumab; Drug: Verteporfin PDT; Drug: Sham Ranibizumab; Drug: Sham verteporfin PDT

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg ranibizumab intravitreal injection
Drug: Verteporfin PDT — Verteporfin (6 mg/m2) intravenous infusion
  Other Names: vPDT
  Arms: Verteporfin PDT
Drug: Sham Ranibizumab — Empty vial to mimic the intravitreal injection
Drug: Sham verteporfin PDT — Sham vPDT intravenous infusion of dextrose 5% solution followed by light application (PDT).

SUMMARY:
This study is designed to evaluate the efficacy and safety of two different dosing regimens of 0.5 mg ranibizumab given as intravitreal injection in comparison to verteporfin PDT in patients with visual impairment due to choroidal neovascularization (CNV) secondary to pathologic myopia (PM).

ELIGIBILITY:
Inclusion Criteria:

* Visual impairment due to choroidal neovascularization (CNV) secondary to PM
* Best corrected visual acuity (BCVA) in the study eye > 24 and < 78 Early Treatment Diabetic Retinopathy Study (ETDRS) letters
* High myopia (> -6D), anterior-posterior elongation > 26 mm; posterior changes compatible with the pathologic myopia
* Either lesion types in the study eye: subfoveal, juxtafoveal, extrafoveal

Exclusion Criteria:

* Patients with uncontrolled systemic or ocular diseases
* Blood pressure > 150/90 mmHg
* History of pan-retinal, focal/grid laser photocoagulation or intraocular treatment with any anti-VEGF or vPDT in the study eye
* Intravitreal treatment with corticosteroids or intraocular surgery within last 3 months in the study eye

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (66):
- Austria (2):
  - Novartis Investigative Site, Vienna, Austria
  - Novartis Investigative Site, Linz, Upper Austria
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- France (5):
  - Novartis Investigative Site, Bordeaux, France
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Regensburg
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- India (5):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, New Delhi, New Delhi
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Bangalore
- Italy (4):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Udine, UD
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
- Novartis Investigative Site, Riga, Latvia
- Lithuania (2):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Novartis Investigative Site, Bielsko-Biala, Poland
- Portugal (2):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Porto
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Etlik / Ankara
- United Kingdom (3):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Ceklic L, Wolf-Schnurrbusch U, Gekkieva M, Wolf S. Visual acuity outcome in RADIANCE study patients with dome-shaped macular features. Ophthalmology. 2014 Nov;121(11):2288-9. doi: 10.1016/j.ophtha.2014.06.012. Epub 2014 Aug 8. No abstract available. PMID 25109929
- [Derived] Wolf S, Balciuniene VJ, Laganovska G, Menchini U, Ohno-Matsui K, Sharma T, Wong TY, Silva R, Pilz S, Gekkieva M; RADIANCE Study Group. RADIANCE: a randomized controlled study of ranibizumab in patients with choroidal neovascularization secondary to pathologic myopia. Ophthalmology. 2014 Mar;121(3):682-92.e2. doi: 10.1016/j.ophtha.2013.10.023. Epub 2013 Dec 8. PMID 24326106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 334 patients screened, 277 patients were randomized into the study on a 2:2:1 basis: 106 patients to Group I (treatment with ranibizumab according to visual acuity stabilization), 116 patients to Group II (ranibizumab treatment according to disease activity), and 55 patients to Group III (treatment with vPDT)
Groups:
- 0.5 mg Ranibizumab Driven by Stabilization Criteria: Participants received ranibizumab on day 1 and month 1. Thereafter they received ranibizumab based on stabilization criteria for visual acuity (VA).
- 0.5mg Ranibizumab Driven by Disease Activity: Participants received active ranibizumab on day 1. Thereafter they received ranibizumab treatment based on disease activity criteria
Period: Overall Study
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Started | 106 | 116 | 55
Completed 3 Months | 105 | 116 | 55
Completed 6 Months | 103 | 116 | 55
Completed | 100 | 112 | 55
Not Completed | 6 | 4 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT | Total
Number analyzed (Participants) | 106 | 116 | 55 | 277
Age, Customized [Number; unit: Participants]
  <45 years | 24 (22.6) | 24 (20.7) | 7 (12.7) | 55
  45 -< 55 years | 27 | 21 | 16 | 64
  55-<65 years | 30 | 34 | 14 | 78
  >=65 | 25 | 37 | 18 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 87 | 40 | 209
  Male | 24 | 29 | 15 | 68

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline to Month 1 Through Month 3 on Visual Acuity of the Study Eye
Description: The Best Corrected Visual Acuity (BCVA) was tested using the Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts at baseline and compared to the average from month 1 to month 3.
Time Frame: Baseline, Month 1 through Month 3
Population: Participants from the Full Analysis Set, included all participants who received at least one dose of study drug, with data available for analysis. Missing data were imputed with Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Letters
  Baseline | 55.4 (13.43) | 55.8 (12.59) | 54.7 (13.84)
  Average Month 1 to month 3 | 66.0 (12.98) | 66.4 (12.28) | 56.9 (14.49)

2. Secondary Outcome: Average Change From Baseline to Month 6 in Visual Acuity of the Study Eye
Description: The Best Corrected Visual Acuity (BCVA) was tested using the Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts at baseline and month 6. The overall BCVA score was calculated using the BCVA worksheet.
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Letters
  Baseline | 55.4 (13.43) | 55.8 (12.59) | 54.7 (13.84)
  Average month 1 to month 6 | 69.2 (12.44) | 68.4 (13.56) | 62.7 (14.65)

3. Secondary Outcome: Average Change From Baseline to Month 1 Through Month 12 in Visual Acuity of the Study Eye
Description: The Best Corrected Visual Acuity (BCVA) was tested using the Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity (VA) testing protocol. VA measurements were taken in a sitting position at an initial test distance of 4 meters using ETDRS charts at baseline and Month 1 through 12
Time Frame: Baseline and Month 1 through Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Letters
  Baseline | 55.4 (13.43) | 55.8 (12.59) | 54.7 (13.84)
  Average Month 1 to Month 12 | 68.3 (12.61) | 68.3 (12.45) | 61.1 (14.86)

4. Secondary Outcome: Percentage of Patients With Best Corrected Visual Acuity (BCVA) ≥10 and ≥15 Letters Gain or Reach 84 Letters at Month 3
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained more than 10 or more than 15 of visual acuity at month 3.
Time Frame: Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Percentage of Patients
  Month 3 >=15 letters | 38.1 | 43.1 | 14.5
  Month 3 >= 10 letters | 61.9 | 65.5 | 27.3

5. Secondary Outcome: Percentage of Patients With Best Corrected Visual Acuity (BCVA) ≥10 and ≥15 Letters Gain or Reach 84 Letters at Month 6 and Month 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained more than 10 or more than 15 letters of visual acuity at month 6 and month 12.
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 0
Percentage of Patients
  Month 6 >=15 letters | 46.7 | 44.8 |
  Month 6 >= 10 letters | 71.4 | 64.7 |
  Month 12 >=15 letters | 53.3 | 51.7 |
  Month 12 >= 10 letters | 69.5 | 69.0 |

6. Secondary Outcome: Percentage of Patients With Best Corrected Visual Acuity (BCVA) ≥10 and ≥15 Letter Loss at Month 3
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. A decreased score indicates worsening in acuity. This outcome assessed the percentage of participants who lost more than 10 or more than 15 of visual acuity at month 3.
Time Frame: Month 3
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Percentage of Patients
  Month 3 >=10 letters | 1.9 | 0.9 | 16.4
  Month 3 >= 15 letters | 1.9 | 0 | 7.4

7. Secondary Outcome: Percentage of Patients With Best Corrected Visual Acuity (BCVA) ≥10 and ≥15 Letter Loss at Month 6 and 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. A decreased score indicates worsening in acuity. This outcome assessed the percentage of participants who lost more than 10 or more than 15 of visual acuity at month 6 and 12.
Time Frame: Months 6 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 0
Percentage of Patients
  Month 6 >=10 letters | 1.9 | 2.6 |
  Month 6 >= 15 letters | 0 | 0.9 |
  Month 12 >=10 letters | 4.8 | 1.7 |
  Month 12 >= 15 letters | 1.9 | 0.9 |

8. Secondary Outcome: Change From Baseline in Central Retinal Thickness of the Study Eye Over Time
Description: Retinal thickness was measured by Central Reading Center using patient's Optical Coherence Tomography (OCT) images provided by investigators.
Time Frame: Baseline, Month 3, Month 6 and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 102 | 110 | 55
Microns
  Baseline (n=102,110, 54) | 349.2 (95.05) | 373.1 (127.44) | 352.5 (101.52)
  Month 3 (n= 102,110,54) | 288.3 (70.14) | 295.6 (71.93) | 340.5 (106.03)
  Month 6 (n= 102,110,55) | 283.1 (67.43) | 298.3 (81.16) | 303.5 (76.81)
  Month 12 (n= 102,110,55) | 282.6 (68.62) | 301.8 (88.16) | 294.3 (83.25)

9. Secondary Outcome: Percentage of Patients With Choroidal Neovascularization (CNV) Leakage in the Study Eye
Description: CNV leakage assessment plus other choroid and retinal disorders were assessed by Central Reading Center using patient's fluorescein angiography and color fundus photography images provided by investigators.
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 105 | 116 | 55
Percentage of Patients
  Baseline-Definite | 96.2 | 93.1 | 100.0
  Baseline- Questionable | 1.0 | 0.0 | 0.0
  Baseline-Absent | 1.0 | 0.9 | 0.0
  Baseline- Other | 1.9 | 6.1 | 0.0
  Month 12-Definite | 21.0 | 19.0 | 29.1
  Month 12- Questionable | 0.0 | 0.0 | 1.8
  Month 12-Absent | 68.6 | 69.8 | 65.5
  Month 12- Other | 0.5 | 11.2 | 3.6

10. Secondary Outcome: Number of Ranibizumab Injections Received Prior to Month 3
Description: In order to describe exposure to the study drug the number of ejections was evaluated
Time Frame: Day 1 and prior to month 3
Population: The Safety Set consisted of all patients who received at least one application of study treatment (ranibizumab [sham] and/or vPDT [sham]) and had at least one post-baseline safety assessment
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Verteporfin PDT
Number analyzed (Participants) | 106 | 118 | 53
injections | 2.5 (0.57) | 1.8 (0.82) | 0.0 (0.00)

11. Secondary Outcome: Number of Ranibizumab Injections Received by Patients Randomized to the Ranibizumab Groups, by Period
Description: Number of ranibizumab injections received by patients randomized to the ranibizumab groups, by period
Time Frame: Day 1 prior to month 6 and prior to month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity
Number analyzed (Participants) | 106 | 118
injections
  Day 1 prior to Month 6 | 3.5 (1.46) | 2.5 (1.56)
  Day 1 prior to month 12 | 4.6 (2.59) | 3.5 (2.92)

12. Secondary Outcome: Number of Ranibizumab Injections Received by Patients Randomized to vPDT With Ranibizumab From Month 3 by Period
Description: Number of ranibizumab injections received by patients randomized to the vPDT with ranibizumab groups, by period.
Time Frame: Month 3 up to month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Verteporfin PDT
Number analyzed (Participants) | 53
injections
  Day 1 up to month 6 (n=34) | 1.9 (0.86)
  Day 1 up to month 12 (n=38) | 3.2 (2.54)

ADVERSE EVENTS:
Description: Two participants who were randomized to Visudyne PDT received 0.5mg Ranibizumab and were followed up in the group "Driven by Disease Activity" therefore, the total of participants at risk in the safety section is discrepant by a number of 2 in each of these groups.
Groups:
- Visudyne PDT: Grp III With 0.5mg Ranibizumab From Month 3: After month 3 participants received active ranibizumab, active vPDT or a combination of the two if needed.
- Visudyne PDT: Grp III Without 0.5mg Ranibizumab From Month 3: After month 3 participants did not receive active ranibizumab
Arm/Group | 0.5 mg Ranibizumab Driven by Stabilization Criteria | 0.5mg Ranibizumab Driven by Disease Activity | Visudyne PDT: Grp III With 0.5mg Ranibizumab From Month 3 | Visudyne PDT: Grp III Without 0.5mg Ranibizumab From Month 3
Serious Adverse Events (participants affected / at risk) | 7/106 | 6/118 | 0/38 | 0/15
Other Adverse Events (participants affected / at risk) | 46/106 | 47/118 | 17/38 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5 mg Ranibizumab Driven by Stabilization Criteria (N=106) | 0.5mg Ranibizumab Driven by Disease Activity (N=118) | Visudyne PDT: Grp III With 0.5mg Ranibizumab From Month 3 (N=38) | Visudyne PDT: Grp III Without 0.5mg Ranibizumab From Month 3 (N=15)
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Corneal erosion (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Retinoschisis (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5 mg Ranibizumab Driven by Stabilization Criteria (N=106) | 0.5mg Ranibizumab Driven by Disease Activity (N=118) | Visudyne PDT: Grp III With 0.5mg Ranibizumab From Month 3 (N=38) | Visudyne PDT: Grp III Without 0.5mg Ranibizumab From Month 3 (N=15)
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Blindness (Study eye) (Eye disorders) | 0 | 0 | 1 | 1
Cataract (Study eye) (Eye disorders) | 1 | 2 | 0 | 1
Conjunctival haemorrhage (Study eye) (Eye disorders) | 12 | 12 | 2 | 0
Conjunctival hyperaemia (Study eye) (Eye disorders) | 1 | 0 | 0 | 1
Conjunctivitis (Fellow eye) (Eye disorders) | 4 | 0 | 0 | 1
Dry eye (Fellow eye) (Eye disorders) | 3 | 3 | 0 | 1
Dry eye (Study eye) (Eye disorders) | 4 | 2 | 0 | 1
Eye pain (Study eye) (Eye disorders) | 4 | 4 | 1 | 1
Ocular hypertension (Fellow eye) (Eye disorders) | 0 | 2 | 1 | 1
Punctate keratitis (Study eye) (Eye disorders) | 8 | 3 | 2 | 0
Visual impairment (Study eye) (Eye disorders) | 0 | 0 | 2 | 0
Vitreous detachment (Study eye) (Eye disorders) | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Injection site haemorrhage (Study eye) (General disorders) | 3 | 3 | 2 | 0
Conjunctivitis viral (Study eye) (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 12 | 12 | 1 | 2
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1
Intraocular pressure increased (Study eye) (Investigations) | 3 | 7 | 4 | 0
Myositis (Study eye) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Headache (Nervous system disorders) | 8 | 11 | 1 | 0
Hypertension (Vascular disorders) | 3 | 5 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.